CLINICAL TRIAL: NCT00276965
Title: Comparing the Safety and Effectiveness of a Mood Stabilizing Medication, an Antidepressant Medication, and a Combination of Both Medications to Treat Symptoms of Bipolar Type II Depression
Brief Title: Bipolar II Depression: Lithium, SSRI, or the Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH074707 (NIH); R01MH074707 (NIH); DATR A5-ETMA
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Disorder; Depression
Keywords: Bipolar II Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Sertraline; Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Participants will take lithium only.
  Interventions: Drug: Lithium carbonate
- B (Experimental): Participants will take lithium and sertraline.
  Interventions: Drug: Sertraline; Drug: Lithium carbonate
- C (Experimental): Participants will take sertraline only.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Sertraline or placebo for sertraline starting at 25 mg per day, up to maximum of 200 mg per day
  Other Names: Zoloft
  Arms: B; C
Drug: Lithium carbonate — Lithium or placebo for lithium starting at 150 mg per day; target dose of 900mg per day. Maximum dose based on clinical response and serum levels (maximum serum level of 1.2 mEq/L).
  Other Names: Eskalith, Lithobid
  Arms: A; B

SUMMARY:
This study will compare the safety and effectiveness of a mood stabilizing medication, an antidepressant medication, and a combination of both medications to treat symptoms of bipolar type II depression.

DETAILED DESCRIPTION:
Bipolar type II depression (BD II) is a less severe type of bipolar disorder. BD II is characterized by one or more depressive episodes and at least one hypomanic episode. During hypomanic episodes, people experience especially energetic or anxious moods, and their thoughts are more sporadic than usual, but they do not experience the severity of mania. Symptoms of BD II are known to impair daily functioning as well as cause distress and even suicide. Antidepressant medication alone is not recommended for people with bipolar disorder because manic symptoms usually worsen. It is unknown whether the same recommendation should apply to people with BD II. Sertraline is a selective serotonin reuptake inhibitor (SSRI) antidepressant that increases levels of serotonin, helping the brain to maintain mental stability. It is often used to treat depression, panic attacks, and other disorders. Lithium is a mood stabilizing medication that decreases abnormal brain activity and is used to treat and prevent recurring episodes of mania in people with bipolar disorders. This study will evaluate the effectiveness of lithium alone, sertraline alone, and lithium with sertraline to treat symptoms of BD II.

Participation in this double-blind study will last up to 18 weeks. Participants will be randomly assigned to receive either lithium, sertraline, or lithium and sertraline. Both medications will initially be given at a low dose and then gradually increased over 2 weeks. For the remainder of the study, dosages will be adjusted as necessary. Study visits will occur every week for the first 6 weeks and then every other week for the remaining 10 weeks. During all study visits, participants will complete a psychiatric assessment and questionnaires about their current mood and any treatment side effects. Urine and blood collection may occur at selected times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for bipolar type II disorder by Structured Clinical Interview for DSM-IV (SCID)
* Meets DSM-IV criteria for current depressive episode
* Inventory of Depressive Symptomology (IDS-C) score greater than 22
* Clinical Global Impression Scale for Bipolar Illness (CGI-BP) depression subscale score greater than 3 (mildly ill or greater) and mania subscale score of 1 (not ill)
* Young Mania Rating Scale (YMRS) score less than 8
* Willing to discontinue antidepressant medication
* Considered stable and does not require adjustments in treatment for other conditions or illnesses
* Willing to use an effective form of birth control throughout the study
* Speaks English

Exclusion Criteria:

* Pregnant or breastfeeding
* Unsuccessfully treated for more than 6 weeks with sertraline or lithium for depression
* Suicidal
* Significant alcohol or substance abuse or dependence within 3 months of study entry
* Diagnosed with Axis II borderline personality disorder
* Psychotic
* Organic mood disorder (e.g., head trauma or cerebrovascular accident preceding mood episode)
* Active hepatitis, liver failure, or kidney failure
* Creatinine greater than 1 mg/dL
* Liver function tests greater than 3 times the upper limit of normal
* Abnormal thyroid-stimulating hormone
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2006-09; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determine switch rate to Mania/hypomania | Measured at week 16

SECONDARY OUTCOMES:
Side effects | Measured at week 16
Antidepressant response | Measured at week 16
Mood variability | Measured at week 16

CONTACTS AND LOCATIONS:
Overall Officials: Lori Altshuler, MD, Principal Investigator — UCLA Mood Disorders Research Program
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Stanford University - Bipolar Research Program, Palo Alto, California
  - Lindner Center of HOPE, affliated with University of Cincinnati Medical Center, Mason, Ohio